CLINICAL TRIAL: NCT06291571
Title: Assessment of Microorganisms and Host Response In Liver Diseases
Acronym: MILD
Status: Not yet recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 324543
Record Dates: First submitted 2024-02-16; First posted 2024-03-04 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Gut Microbiome; Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Liver diseases: Patients with documented liver diseases
- Control: Healthy volunteers without evidence of liver disease

SUMMARY:
The normal human gut is home to millions of microbes including bacteria, fungi, and viruses, collectively forming the gut microbiota, which exists in harmony within us. Much research is still required to fully understand the contribution of microbes resident in the large intestine in liver diseases. The liver receives blood from the gut carrying all the necessary nutrients needed for our body but also has to deal with toxins derived from the microbes residing in the intestines. The gut microbiota is altered in liver disease. We still do not know clearly how this change impacts liver function and the health of liver patients. The purpose of our study is to answer this question by assessing the gut microbiota using modern microbiological and molecular methods. By studying the alterations in the gut microbiota in patients with liver disease we can understand how they affect our immune system and metabolism. This will help design novel medicinal products to prevent and treat liver disease.

DETAILED DESCRIPTION:
Purpose and design:

The key question of this research study is to elucidate the role of the gut microbiota (bacteria, fungi and viruses) in the development and progression of liver disease. There is a large amount of existing literature which suggests that there is a change in the nature of the gut microbes in liver diseases. However, the specific role of the 'gut virome' in liver disease is still an emerging field. Its relationship with the bacteria and fungi in the lumen and interaction with the host immune system needs to be characterised in liver diseases. This study aims to look at the host-microbe dynamics in liver diseases, which will not only lead to a better understanding of the pathogenesis of these diseases but also help in designing therapeutic interventions to prevent progression. The proposal has been peer-reviewed by colleagues at Aberdeen Royal Infirmary. Wider dissemination of the results will be done through publications in scientific journals and through public engagement forums.

Recruitment:

Patients will be recruited from the Peter Brunt Gastrointestinal (GI) and Liver clinic, and the GI and liver ward at Aberdeen Royal Infirmary. Outpatient attendees will be sent participant information sheets by mail before their clinical attendance along with their clinic appointment letter, for them to have enough time to understand the information. At their clinic appointment, they will be consented by a member of the clinical team, and a collection kit handed to them for a faecal sample. For patients with liver disease receiving treatment on the ward, we will collect faecal samples after informed consent is obtained. Information regarding the cause and stage of liver disease will be routinely collected from the case records of these patients. We would also like to obtain faecal samples from a subgroup of patients over a longer time course to see the evolution of gut microbiota over time. We will request two more faecal samples over a period of six months. All the necessary collection containers and information for delivery of these samples to the research laboratory at the Institute of Medical Sciences, University of Aberdeen will be provided. Finally, we may request a blood sample from a subset of patients (n=25) for challenge studies. A total of 30 ml of blood will be collected from this subgroup of patients. These patients will be consented specifically by the clinical team.

A very small group of patients will be identified when they are listed for a liver biopsy. This procedure is done for diagnostic reasons or to stage the disease in a specific cohort of patients with liver disease. The decision to do the biopsy is taken by their consultant hepatologist. The biopsy is done in a day-case unit in a planned manner. The patients are sent an appointment letter to come in for the procedure. The participation information sheets will be sent along with these letters, to consider the information in advance. They will be consented by a member of the clinical team on the day of the biopsy.

The liver biopsy is performed by a consultant radiologist. A portion of liver tissue in excess of that required for diagnostic purposes will be cut off from the main sample. The portion will not be more than 0.5 cm with at least 2 cm of liver tissue sent to the labs for clinical and pathological assessment. The portion taken for research will be kept and transported to the University of Aberdeen lab in a liquid nitrogen flask for work package 3 assessment. Cells will then be isolated from these samples for single-cell RNA sequencing analysis (ScRNAseq) analysis. Liver tissue will also be utilised to perform spatial transcriptomics which will localise the exact area of metabolic alteration. These cells will also be used to create tissue organoids.

There are two liver research nurses and a Hepatology research fellow who will help in co-ordinating the study. There are five consultant hepatologists and specialist registrars who will help in identifying prospective patients. We would anticipate the collection of 200 liver disease patient sample sets and a corresponding number of appropriately matched control subjects over the five-year proposed study period for the wider study. We would anticipate 50 subjects for the liver biopsy sub-group study in the same time period.

Control subjects will be healthy volunteers recruited from the University of Aberdeen and Aberdeen Royal Infirmary. The study will be advertised through pamphlets. The control participants will be contacted by the research team and will be given the participation information sheets which will be sent by email or handed over in person, 24 hours before consent is obtained. This will ensure they have time to read and understand the research study. An initial screening meeting will take place during which the volunteer will meet a member of the research team. They will be asked to complete a basic health questionnaire detailing age, weight and details of any relevant health conditions and regular medication to ensure that they meet the inclusion/exclusion criteria for the study. If they meet the inclusion criteria, then they will be asked to sign a consent form and will then be formally recruited into the study. They will be given a study number that will be used at all times to keep their identity anonymous.

A subject log will be maintained for all the patients and controls recruited in the study which will be kept securely in a locked cabinet in the University of Aberdeen.

Methodology

The study will be carried out in the University of Aberdeen, Institute of Medical Sciences and Rowett Institute research laboratories. The study aims to elucidate the role of the gut microbiota and host immune response in liver disease through three work packages as described below:

Work package 1: Investigation of the alteration of gut microbiota in liver diseases

This work package involves collection of faecal samples from eligible patients and healthy controls for the following assessments:

A) To investigate the alteration of the gut microbiota in patients with liver diseases: Molecular analyses will require DNA and RNA extraction from faecal samples collected from patients. PCR based assessment will be employed using both universal and also group/species directed approaches to study microbial diversity. Following PCR analysis, other analytical methods may be employed including (but not exclusively) clone library construction and Sanger sequencing and also probing based approaches. Omics based approaches like 16sRNA gene sequencing, metagenomics, metatranscriptomics, metabolomics and metaproteomics will also be used to study microbial diversity and function.

B) Isolate and characterise the pathogenic potential of specific microbes which are associated with liver diseases: Microbiological assessment of faecal samples will allow us to enumerate specific microbes (bacteria, viruses, and fungi) from samples using conventional microbiology culture techniques. These isolates will then be identified and assessed for their pathogenetic potential. This will involve genomic assessment of pathogenicity utilising techniques like whole genome sequencing to characterise specific traits. We will also perform metabolomic assessment of pathogenic microbes to look for alteration in pathways pertaining to bile salt, alcohol, and short chain fatty acid metabolism. This will involve transcriptomic assessment of the pathogenic strains as well as gas chromatography to study the by-products of their metabolism.

Work package 2: Assessment of host response to specific microbes in liver diseases This work package will involve collection of 30 ml of blood from patients and controls. This group of subjects will be consented specifically for blood testing. This blood will be used to generate macrophages which will be needed for the challenge studies. Pathogenic microbes identified in Study 1 will be assessed for their pro-inflammatory potential through challenge experiments on cell lines, tissue organoids and experimental animal models. Blood taken at the time of recruitment will be assessed for evidence of inflammatory mediators following challenge with infectious agents identified in Study 1. Whole blood collected ~ 30 ml (2 tablespoons) will have a panel of bacterial/viral and fungal cells added and these will be incubated for up to 48 hours. Evidence of inflammatory development will be studied using molecular techniques including (but not exclusively) ELISA and flow cytometric analysis. In a proportion of subjects, blood will be taken to extract peripheral blood monocyte cells (PBMCs) to assess the systemic immune response against these putative pathogens.

Work package 3: Characterise the changes in the liver immune microenvironment by analysing liver biopsies from patients. This work package will be done to elucidate the inflammatory changes that are occurring within the liver in response to the gut pathogens. A small subgroup of patients who are undergoing liver biopsy for clinical reasons will be consented for a small portion of liver tissue in excess of what is required for diagnostic purposes. The larger portion will be sent off for pathological assessment. This small excess portion will be cut off from the liver biopsy by the radiologist and handed over immediately to a member of the research team. This will be transported in a liquid nitrogen flask to the University of Aberdeen lab for processing. Hepatocytes will then be isolated from these liver biopsy samples for single-cell RNA sequencing analysis (ScRNAseq). Liver tissue will also be utilized to perform spatial transcriptomics which will localize the exact area of metabolic alteration.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent
2. Definitive diagnosis of specific liver disease utilising clinical, biochemical, and radiological tests
3. Male or female aged between 18-70 years
4. Able to understand written or verbal information in English

Exclusion Criteria:

1. Pregnancy and breastfeeding
2. Treatment with antibiotics in the last month
3. Treatment with steroids or immunosuppressive drugs in the last month
4. Regular consumption of over-the-counter prebiotics and probiotics from pharmacies or other retailers in the last month.
5. Known gastrointestinal disease, including but not limited to ulcerative colitis, Crohn's disease, coeliac disease, microscopic colitis, diverticulitis, irritable bowel syndrome
6. Patients diagnosed with cancer who are on chemotherapy, radiotherapy, or immunotherapy within the last 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in clinics and wards in secondary care.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2029-02-28 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
To identify the bacterial, fungal, and virological agents present in patients with liver disease as opposed to controls | 5 years
  Microbiome analysis in liver patients and controls

SECONDARY OUTCOMES:
To assess the host immune response against specific microbes isolated from patients with liver disease and controls | 5 years
  Immune response in liver patients and controls
To characterise the changes in the liver immune microenvironment by analysing liver biopsies from patients | 5 years
  Liver biopsy analysis

CONTACTS AND LOCATIONS:
Overall Officials: Indrani Mukhopadhya, Principal Investigator — Principal Investigator

IPD SHARING:
Plan to Share IPD: Undecided